CLINICAL TRIAL: NCT04400942
Title: A Retrospective Study for Developing a Nomogram for Predicting Change of Complete Myoma Resection During Hysteroscopic Myomectomy
Brief Title: Predictive Factors for Complete Myoma Resection During Hysteroscopic Myomectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Fabio Barra, Principal Investigator, Ospedale Policlinico San Martino
Other Study IDs: NOM-MYOMA RES
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Uterine Fibroids; Uterine Myomas
MeSH Terms: conditions — Leiomyoma | interventions — Immunologic Memory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with uterine myomas undergoing hysteroscopic myomectomy
  Interventions: Diagnostic Test: Transvaginal ultrasound; Behavioral: Anamnesis; Procedure: Operative hysteroscopy

INTERVENTIONS:
Diagnostic Test: Transvaginal ultrasound — Transvaginal ultrasonographic scan aims to evaluate number, size (diameter and volume), location and appearance of submucous uterine myomas, concomitant presence of adenomyosis
Behavioral: Anamnesis — Anamnesis aims to collect data about age, BMI, previous hormonal therapies (such as ulipristal acetate or gonadotropin-releasing hormone agonists) with submucous uterine myomas
Procedure: Operative hysteroscopy — Operative hysteroscopy allows a direct evaluation of number, size (diameter and volume), location and appearance of submucous uterine myomas. This exam allows the resection of the myomas.

SUMMARY:
The aim of this observational retrospective analysis is to evaluate predictive factors for complete myoma resection during hysteroscopic myomectomy for developing and validating a nomogram.

This tool can help clinicians to support the patient in making an informed decision about therapeutic options for uterine submucous myomas by defining risk factors predicting a high complexity myomectomy.

DETAILED DESCRIPTION:
Overall, 10% of all uterine myomas are submucosal. These myomas spread into the uterine cavity, lifting the endometrial mucosa, and are a common cause of abnormal uterine bleeding, dysmenorrhea, early miscarriage and they may be a cause of infertility.

Hysteroscopic myomectomy is the surgical procedure of choice for the treatment of submucosal myomas, because it is minimally invasive and has the advantage of preserving the integrity of the uterine wall.

The characteristics of the myomas (size, number and location) enables the surgeon to choose the surgical approach that will provide the best outcome for the patient, and may predict the chances of a complete hysteroscopic resection of myomas in one procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients with ultrasonographic diagnosis of uterine myomas

Exclusion Criteria:

* patients with previous incomplete hysteroscopic myoma resection;
* patients undergoing additional surgical procedures performed by hysteroscopy (such as, resection of endometrial polyps);
* patients undergoing associated non-hysteroscopic surgical procedures;
* patients with severe cardiovascular disease, decompensated diabetes and severe hematologic disorders

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with trasonographic diagnosis of uterine myomas undergoing hysteroscopic myomectomy
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with complete resection of myomas | At the end of the hysteroscopic procedure

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genoa, Italy

REFERENCES:
- [Background] Vargas MV, Moawad GN, Sievers C, Opoku-Anane J, Marfori CQ, Tyan P, Robinson JK. Feasibility, Safety, and Prediction of Complications for Minimally Invasive Myomectomy in Women With Large and Numerous Myomata. J Minim Invasive Gynecol. 2017 Feb;24(2):315-322. doi: 10.1016/j.jmig.2016.11.014. Epub 2016 Dec 7. PMID 27939896
- [Background] Ferrero S, Tafi E, Racca A, Leone R, Maggiore U, Remorgida V, Venturini PL. Ulipristal Acetate Prior to High Complexity Hysteroscopic Myomectomy: Prospective Study. J Minim Invasive Gynecol. 2015 Nov-Dec;22(6S):S181. doi: 10.1016/j.jmig.2015.08.666. Epub 2015 Oct 15. No abstract available. PMID 27678974